CLINICAL TRIAL: NCT04408014
Title: Seroepidemiological Study of SARS-CoV-2 Infection in Population Subgroups in the State of São Paulo
Brief Title: Seroepidemiological Study of SARS-CoV-2 (COVID-19) Infection in Population Subgroups in the State of São Paulo
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVID-19-Epi-01
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: COVID; SARS-CoV 2
MeSH Terms: interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasopharyngeal Swab, Oropharyngeal Swab and Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- HC-USP: Home contacts of health professionals diagnosed with COVID-19 at the Hospital of Clínic of Medicine School of the University of São Paulo
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab
- CORAS: Refugees living in the city of São Paulo
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab
- Hemocenter: Blood Donors of the Pró-Sangue Hemocenter Foundation of São Paulo
  Interventions: Diagnostic Test: Serological test
- CPP - Butantan Penitentiary Progression Center: Participants of the CPP - Butantan Penitentiary Progression Center
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab
- CHSP - Penitentiary System Hospital Center: Participants of the CHSP - Penitentiary System Hospital Center
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab
- SABE (Health, Wellness and Aging): Participants of the SABE Project (Health, Wellness and Aging)
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab
- ILPI - Long-Term Care Institution for the Elderly: Residents of the Long-Term Care Institution for the Elderly of Botucatu
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab
- ICR-USP - Children's Institute of HCFMUSP: Home contacts of children and adolescents diagnosed with COVID-19, attended at the Children's Institute of HCFMUSP
  Interventions: Diagnostic Test: Serological test; Diagnostic Test: Nasopharyngeal Swab; Diagnostic Test: Oropharyngeal Swab

INTERVENTIONS:
Diagnostic Test: Serological test — IgM and IgG for SARS-CoV-2
Diagnostic Test: Nasopharyngeal Swab — PCR for SARS-CoV-2
  Groups: CHSP - Penitentiary System Hospital Center; CORAS; CPP - Butantan Penitentiary Progression Center; HC-USP; ICR-USP - Children's Institute of HCFMUSP; ILPI - Long-Term Care Institution for the Elderly; SABE (Health, Wellness and Aging)
Diagnostic Test: Oropharyngeal Swab — PCR for SARS-CoV-2
  Groups: CHSP - Penitentiary System Hospital Center; CORAS; CPP - Butantan Penitentiary Progression Center; HC-USP; ICR-USP - Children's Institute of HCFMUSP; ILPI - Long-Term Care Institution for the Elderly; SABE (Health, Wellness and Aging)

SUMMARY:
Seroepidemiological Study of SARS-CoV-2 Infection in Population Subgroups in the State of São Paulo

DETAILED DESCRIPTION:
This is a cross-sectional study to estimate the prevalence of antibodies against SARS-CoV-2 is different population subgroups in the State of São Paulo

ELIGIBILITY:
Inclusion Criteria:

* All potential volunteers invited to participate in the study.

Exclusion Criteria:

* All potential eligible participants, but who do not show interest in participating in the study.

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Home contacts of health professionals at the Hospital das Clínicas of the Medical School of USP diagnosed with COVID-19;
  * Refugees living in the city of São Paulo - CORAS-BR Project;
  * Blood Donors of the Fundação Pró-Sangue Hemocentro de São Paulo
  * Butantan Penitentiary Progression Center participants;
  * Penitentiary System Hospital Center (CHSP) participants;
  * SABE Project - Cohort of the Elderly in the city of São Paulo and their home contacts;
  * Residents of the Long Term Care Institution (ILPI) of Botucatu;
  * Home contacts of children and adolescents with a positive diagnosis for COVID-19, attended at Instituto da Criança, HCFMUSP.
Sampling Method: Probability Sample
Enrollment: 18901 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of antibodies against SARS-CoV-2 through serological testing | 1 month
  IgM and IgG antibodies against SARS-CoV-2
Frequency of participants with a positive RT-PCR test result for SARS-CoV-2 | 1 month
  Positive RT-PCR test result for SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Precioso, MD, PhD, Study Chair — Instituto butantan
Locations (1):
- Avenida Vital Brasil 1500, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No